CLINICAL TRIAL: NCT05606029
Title: A Case Series On Incidentally Detected Gallbladder Malignancy
Status: Completed | Type: Observational
Sponsor: Osmania Medical College (Other Government)
Responsible Party: Principal Investigator, Dr. Sathaiah Dadi, MS General Surgery, Principal investigator, Osmania Medical College
Other Study IDs: SOUMY2345
Record Dates: First submitted 2022-10-25; First posted 2022-11-04 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Gallbladder Malignant Neoplasm
Keywords: Gallbladder,; Polyp; Gallstones; Malignancy; Perforation
MeSH Terms: conditions — Gallbladder Neoplasms; Polyps; Gallstones; Neoplasms | interventions — Cholecystectomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who underwent cholecystectomy for benign conditions: In those who underwent cholecystectomy for benign conditions, the histopathological analysis showed the malignancy.
  Interventions: Procedure: Cholecystectomy, extended cholecystectomy

INTERVENTIONS:
Procedure: Cholecystectomy, extended cholecystectomy — Cholecystectomy and histopathological evaluation
  Other Names: Histopathological evaluation of the specimen

SUMMARY:
A retrospective analysis of data, using the Hospital records of all the patients who underwent cholecystectomy for benign conditions at Osmania General Hospital in a year (2019).

DETAILED DESCRIPTION:
A retrospective analysis of hospital records of patients who underwent Cholecystectomy in a year duration (2019) for any benign condition, diagnosed and confirmed histopathologically as Gallbladder Malignancy.

There are a total of one hundred and eighty patients who underwent cholecystectomy at our hospital (Osmania General Hospital) in 2019, out of which seven patients' histopathological diagnosis was gall bladder malignancy. We reviewed all the case's history, cross-checked the histopathological slides, and confirmed the diagnosis. To avoid the bias of covid-19 pandemic in surgical practice we confined the patient records to the pre-pandemic period of one-year duration (2019).

A total of 180 patients underwent cholecystectomy for various benign conditions in one year, out of which seven patients confirmed histopathologically with Gallbladder malignancy.

Total no of patients : 180 Diagnosed with malignancy : 7 percentage 3.8%

Among these seven, three patients converted from laparoscopic to open procedure for difficulty with resection, two patients are posted for surgery considering empyema of gall bladder preoperatively, one patient in view of gall bladder perforation, and for two patients preoperative diagnosis was gall bladder polyp.

Converted from Lap to Open: 3 Pre-op GB Polyp : 2 Perforated GB : 1 Empyema GB : 2

Only one patient is 40 years old and others are more than 50 years, and two of them are males.

Total : 7 100% Males : 2 28.5% Females : 5 71.5%

Out of a total of 180 patients who underwent cholecystectomy, 117 are females and 63 are males

Total : 180 Males : 63 Females : 117

Out of 180, the age distribution is as follows

Age. Percentage 20 - 29 0 30 - 39 0 40 - 49 0.005 >50. 99.99

It implies that the malignancy rate increases with an increase in the patient's age more than 50years and also with gender (Females > males).

ELIGIBILITY:
Inclusion Criteria: All patients who underwent cholecystectomy for benign conditions -

Exclusion Criteria: All those who already diagnosed with gallbladder malignancy

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the patients who underwent cholecystectomy for benign conditions like gall stones, polyps,. Etc,.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Diagnosed with Gallbladder malignancy | For one year
  Those who underwent cholecystectomy for benign conditions are diagnosed with gallbladder malignancy

CONTACTS AND LOCATIONS:
Overall Officials: Sathaiah Dadi, MS Gen Surg, Principal Investigator — Osmania Medical College
Locations (1):
- Osmania General Hospital, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-08): https://cdn.clinicaltrials.gov/large-docs/29/NCT05606029/Prot_SAP_000.pdf